CLINICAL TRIAL: NCT00369798
Title: Antidepressant Effects on cAMP Specific Phosphodiesterase (PDE 4) in Depressed Patients
Brief Title: Antidepressant Effects on cAMP Specific Phosphodiesterase (PDE4) in Depressed Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060215; 06-M-0215
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-10-12

CONDITIONS: Major Depressive Disorder; Healthy
Keywords: Unipolar Depression; Phosphorylation; Affinity States; Compartment Analysis; (R)-(11)C Rolipram; Depression; Major Depressive Disorder; MDD; Healthy Volunteer; HV
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression | interventions — Magnetic Resonance Spectroscopy; Rolipram

INTERVENTIONS:
Procedure: PET scan
Drug: Rolipram

SUMMARY:
The primary purpose of this protocol is to compare PDE4 levels before and after starting a selective serotonin reuptake inhibitor (SSRI) sertraline, citalopram or escitalopram in unmedicated depressed patients. The secondary purpose is to compare PDE4 levels between unmedicated depressed patients and healthy subjects.

DETAILED DESCRIPTION:
Although direct pharmacological effects of antidepressant should manifest rapidly, before significant symptom relief appears, typically antidepressant treatment needs to be continued for 2 to 4 weeks. This delayed onset of clinical effects indicates involvement of adaptive changes in antidepressant effects. Rodent studies have consistently shown upregulation of the 3, 5-cyclic adenosine monophosphate (cAMP) system induced by different types of chronic but not acute antidepressant treatment including serotonin and norepinephrine uptake inhibitors, monoamine oxidase inhibitors, tricyclic antidepressants, lithium and electroconvulsions. cAMP is synthesized from adenosine 5-triphosphate (ATP) by adenylyl cyclase and metabolized by cyclic nucleotide phosphodiesterases (PDEs). Type 4 PDE (PDE4) is selective to cAMP in the brain. Among components of the cAMP pathway, PDE4 appears to be critical for antidepressant effects because an inhibitor of PDE4, 4-[3-(cyclopenotoxyl)-4-methoxyphenyl]-2-pyrrolidone (rolipram), showed antidepressant effects both in animals and humans, and various forms of antidepressant treatment induced increase in PDE4 in rodents. However, without imaging the cAMP pathway before and after antidepressant treatment in depressives, it is not possible to study adaptive changes in the signal transduction system and its role in the symptom relief.

Recently (R)-[(11)C]rolipram has been successfully used to image PDE4 in animals and humans. We have confirmed that PDE4 levels can be measured reliably by performing (R)-[(11)C]rolipram positron emission tomography (PET) with multiple arterial sampling even in rats. The primary purpose of this protocol is to compare PDE4 levels before and after starting a selective serotonin reuptake inhibitor (SSRI) sertraline, citalopram or escitalopram in unmedicated depressed patients. The secondary purpose is to compare PDE4 levels between unmedicated depressed patients and healthy subjects. Baseline scans of patients will be used for this second comparison. For the first time, these comparisons have become possible with the new PET agent (R)-[(11)C]rolipram. The findings will advance understanding on the role of cAMP signal transduction system in the pathology of depression and the mechanisms of antidepressant effects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Volunteers (n = 70)

Healthy Control Sample (n = 70): Sixty of these volunteers will have brain PET scans and 10 of these have only blood sampling to compare (R)-[(11)C]rolipram levels in artery and vein. Healthy subjects (ages 18-55) will be selected who have not met criteria for any major psychiatric disorder, have no known first-degree relatives with mood disorders, and have a current score on the Hamilton Depression Rating Scale (HDRS; 17 item) (Williams 1988) in the not depressed range (less than or equal to 7). Control subjects will be matched to depressed subjects for age and gender. Forty of these subjects will have (R)-[(11)C]rolipram PET scans with blood sampling and 10 subjects have only blood sampling without PET scan. The healthy volunteers who are used to measure the difference in (R)-[(11)C]rolipram concentration between the artery and the vein will not undergo psychiatric assessment because the data will not be compared with those of patients.

MDD Samples (n = 65)

MDD Sample-Currently Depressed (n = 65): Patients (ages 18-55) will be selected with primary MDD currently depressed by DSM-IV criteria for recurrent MDD and current 17-item HDRS score greater than or equal to 18 or Montgomery-Asberg Depression Rating Scale (MADRS) (Noble et al 1991) greater than or equal to 20 indicating the moderately-to-severely depressed symptoms. All subjects must be physically healthy and aged 18 55 years.

EXCLUSION CRITERIA:

Subjects will be recruited who are drug-na(SqrRoot) ve or who have not received psychotropic drugs for at least 2 weeks (6 weeks for fluoxetine) prior to scanning. Effective medications will not be discontinued for the purposes of the study.

Subjects will also be excluded if they have:

1. serious suicidal ideation or behavior
2. psychosis
3. medical conditions or concomitant medications that are likely to influence PET measurement or have significant interactions with sertraline, citalopram or escitalopram.
4. a history of drug or alcohol abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM-IV criteria)
5. positive urine drug screen
6. current pregnancy (as documented by pregnancy testing prior to scanning)
7. general MRI exclusion criteria
8. major depression that arose following another major medical or psychiatric condition, and
9. prior participation in other research protocols within a year such that radiation exposure would exceed the annual guidelines

For patients who have two [C-11]rolipram PET scans, one before and another after SSRI treatment, previous failures of or intolerance to SSRI may not allow for treatment in the current protocol. In clinical practice, medication can be switched between sertraline and citalopram/escitalopram because sertraline and citalopram/escitalopram have somewhat different therapeutic effects and adverse reactions. Along these lines, we will consider citalopram and its enantiomer escitalopram as being equivalent to each other. Patients will therefore be excluded from the study with two [C-11]rolipram PET scans if they previously failed to respond to adequate treatment trials of all medications available for use in the study, or if they have a history of being unable to tolerate all of the study medications. Specifically, patients will be excluded from the study with two [C-11]rolipram PET scans if they:

j) previously proved unresponsive to therapeutic trials of both sertraline and citalopram/escitalopram.

k) previously developed allergic reactions to both sertraline and citalopram/escitalopram, or discontinued both sertraline and citalopram/escitalopram due to an adverse effect

l) through any combination of therapeutic unresponsiveness and adverse medication effects, are unsuitable for treatment with both sertraline and citalopram/escitalopram

m) prolonged QTc in ECG

Please note that the exclusion criteria j, k, and l do not apply to patients who have one [C-11]rolipram PET without having antidepressant treatment in this protocol.

Additional exclusion criteria applied to control subjects are:

n) subjects with a current or past history of other axis I psychiatric conditions

o) subjects with first-degree family members with current or past history of mood disorder.

Please note that these exclusion criteria (with the exception of f and i) do not apply to the healthy volunteers who are used to measure the difference in (R)-[(11)C]rolipram concentration between the artery and the vein, without PET scanning.

Subjects beyond age 55 are excluded to reduce the biological heterogeneity encompassed by the MDD criteria, and to reduce the variability of PET data.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-08-02; Primary Completion 2016-06-16 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
PET measurement of PDE4 levels. | 3 years

SECONDARY OUTCOMES:
Correlation between PDE4 levels and depression symptoms | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Andersen PH, Klysner R, Geisler A. Cyclic AMP phosphodiesterase activity in rat brain following chronic treatment with lithium, imipramine, reserpine, and combinations of lithium with imipramine or reserpine. Acta Pharmacol Toxicol (Copenh). 1983 Oct;53(4):337-43. doi: 10.1111/j.1600-0773.1983.tb03432.x. PMID 6316725
- [Background] Blier P, de Montigny C. Current advances and trends in the treatment of depression. Trends Pharmacol Sci. 1994 Jul;15(7):220-6. doi: 10.1016/0165-6147(94)90315-8. PMID 7940983
- [Background] Conti M, Nemoz G, Sette C, Vicini E. Recent progress in understanding the hormonal regulation of phosphodiesterases. Endocr Rev. 1995 Jun;16(3):370-89. doi: 10.1210/edrv-16-3-370. No abstract available. PMID 7671852
- [Derived] Fujita M, Richards EM, Niciu MJ, Ionescu DF, Zoghbi SS, Hong J, Telu S, Hines CS, Pike VW, Zarate CA, Innis RB. cAMP signaling in brain is decreased in unmedicated depressed patients and increased by treatment with a selective serotonin reuptake inhibitor. Mol Psychiatry. 2017 May;22(5):754-759. doi: 10.1038/mp.2016.171. Epub 2016 Oct 11. PMID 27725657